CLINICAL TRIAL: NCT04986293
Title: Continuous and Bi-level Positive Airway Pressure for Motion Mitigation of Intra-thoracic Tumors Treated With Radiotherapy
Brief Title: CPAP or BiPAP for Motion Mitigation During Radiotherapy
Acronym: SISTER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, R. Wijsman, Principal Investigator, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL71871.042.19/RT2019-17
Record Dates: First submitted 2021-07-01; First posted 2021-08-02 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Radiotherapy Side Effect; NSCLC; Esophageal Cancer; Malignant Lymphoma
Keywords: BiPAP; CPAP; Mechanical ventilation
MeSH Terms: conditions — Radiation Injuries; Esophageal Neoplasms; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CPAP — Different settings of CPAP and BiPAP will be tested using a home mechanical ventilator
  Other Names: BiPAP

SUMMARY:
When using highly conformal radiotherapy techniques, such as proton therapy, a controlled breathing pattern and a minimal breathing amplitude could greatly benefit the treatment of mobile tumors. This reduction in tumor motion may be achieved with the use of a ventilator that is able to regulate and modulate the breathing pattern. CPAP provides a constant level of positive airway pressure. Compared to spontaneous breathing, the use of CPAP increased lung volume and can result in a significant decrease in tumor movement and a significant decrease in both mean lung and mean heart radiation dose. These results were found in patients treated for limited stage disease, it is not clear if this approach is feasible for patients with more advanced stage of disease that undergo radiotherapy with curative intent.

With Bilevel Positive Airway Pressure (BiPAP), tidal volume excursions are determined by the pressure difference between the set inspiratory positive airway pressure (IPAP) and the set expiratory positive airway pressure (EPAP). This mode of ventilation increases lung volume comparable to CPAP, but also to control tidal volumes and breathing frequency. However, BiPAP has never been studied in the setting of motion mitigation during radiotherapy and BiPAP might be more difficult to adjust to for patients compared to CPAP. Therefore, the current study is proposed to evaluate whether or not CPAP or BiPAP is of benefit in patients that undergo radiotherapy for larger intra-thoracic tumor volumes.

DETAILED DESCRIPTION:
The study will follow a 2-step approach.

First (Phase 1, n=10), the feasibility of short-term use of CPAP and BiPAP and its effects on (regional) lung volumes, tidal volumes and breathing frequency will be investigated in patients with intra-thoracic tumors who are planned for radiotherapy. This is necessary to select the best setting of CPAP or BiPAP with which minimal tumor motion is expected (and that is feasible for the patient).

In the second phase (n=21), the particular setting found in fase 1 is investigated: weekly repeated radiotherapy planning (4D) CT scans with and without CPAP/BiPAP will be aquired to evaluate the influence on tumor motion and dose to the target and organs at risk. Radiotherapy will be deliverd according to local protocol without the use of CPAP/BiPAP.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Stage III/IV (N)SCLC, esophageal cancer or malignant lymphoma that will be treated with curative intent
* WHO 0-2.
* Written informed consent

Exclusion Criteria:

* Facial deformations so that facial mask is impossible to fit
* Noncompliance with any of the inclusion criteria.
* Planned for radiotherapy with fraction dose ≥3 Gy.
* Severe heart failure (LVEF<30%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Lung volume changes induced by the use of mechanical ventilation | 2-3 hours of measurement (only once)
  The primary objective is to evaluate the lung volume changes (in cm3) induced by the use of mechanical ventilation

SECONDARY OUTCOMES:
Feasibility of mechanical ventilation | once every week up to a maximum of 5 consecutive weeks (depending on the duration of the course of radiotherapy)
  Feasibility is expressed as a score (using a Visual Analoge Scale)
Feasibility of mechanical ventilation | once every week up to a maximum of 5 consecutive weeks (depending on the duration of the course of radiotherapy)
  Feasibility is expressed as the duration (minutes) the participant can undergo mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Robin Wijsman, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No